CLINICAL TRIAL: NCT05114603
Title: An Open-label, Multicenter Phase II Clinical Study to Evaluate Safety, Efficacy and PK of HLX208 for Advanced Melanoma With BRAF V600 Mutation
Brief Title: A Phase II Clinical Trial to Evaluate HLX208 in Advanced Melanoma Patients With BRAF V600 Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLX208-MEL201
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2021-10

CONDITIONS: Advanced Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-escalation stage (Experimental): Iinvestigate the safety and determine the MTD of HLX208. Two dose levels of 600mg and 900 mg are planned for dose finding.
  Interventions: Drug: HLX208
- Dose-expansion stage (Experimental): Patients with advanced melanoma will be enrolled in two expansion cohorts, at doses equal to or lower than the MTD, to better characterize the safety, tolerability, PK variability, and preliminary efficacy of single-agent HLX208.
  Interventions: Drug: HLX208

INTERVENTIONS:
Drug: HLX208 — level 1:600mg po Bid level 2:900mg po Bid

SUMMARY:
An open-label, multicenter phase II clinical study to evaluate safety, efficacy and PK of HLX208 for advanced melanoma with BRAF V600 mutation

ELIGIBILITY:
Inclusion Criteria:

* Age>=18Y
* Good Organ Function
* Expected survival time ≥ 3 months
* advanced melanoma with BRAF V600 mutation that have been diagnosed
* ECOG score 0-1;

Exclusion Criteria:

* Previous treatment with BRAF inhibitors or MEK inhibitors
* Symptomatic brain or meningeal metastases (unless the patient has beenon > treatment for 3 months, has no evidence of progress on imagingwithin 4 weeks prior to initial administration, and tumor-related clinicalsymptoms are stable).
* Severe active infections requiring systemic anti-infective therapy
* A history of other malignancies within two years, except for cured carcinoma in situ of the cervix or basal cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
ORR | from first dose to the last patient was followed up for 6 month
  Objective response rate(assessed by independent radiological review committee (IRRC) based on the e RECIST Version 1.1)

SECONDARY OUTCOMES:
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier)，assessed up to 1 years
  Progression-free survival(PFS):assessed by IRRC and the investigator based on the RECIST Version 1.1
DOR | from the first occurrence of a documented CR or PR (whichever recorded earlier) to the time of first documented disease progression or death (whichever occurs first) assessed up to 1 years
  Duration of response
OS | from the first dose to the time of death due to any cause，assessed up to 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Peking University Cancer Hospita, Beijing, Beijing Municipality
  - Hunan cancer hospital, Changsha
  - West China Hospital of Sichuan University, Chendu
  - Fujian cancer hospital, Fujian
  - Shangxi Bethune Hospita, Taiyuan
  - union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Henan cancer hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No